CLINICAL TRIAL: NCT01637298
Title: The Thai Red Cross AIDS Research Centre
Brief Title: Biomarkers to Detect Anal Intraepithelial Neoplasia in Thai Men Who Have Sex With Men
Status: Completed | Type: Observational
Sponsor: Thai Red Cross AIDS Research Centre (Other)
Collaborators: University of California, San Francisco (Other); SEARCH Research Foundation (Other); Chulalongkorn University (Other)
Responsible Party: Sponsor
Other Study IDs: AIN Study
Record Dates: First submitted 2012-07-02; First posted 2012-07-11 (Estimated); Last update posted 2017-05-09 (Actual); Status verified 2017-05

CONDITIONS: Anal Intraepithelial Neoplasia
Keywords: Histological HGAIN; detected biomarkers; MSM population; HPV subtypes; AIN study; HIV-positive and HIV-negative MSM; anal cytology and biomarkers; likelihood of AIN development at month 12 and yearly thereafter
MeSH Terms: conditions — HIV Seropositivity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The goals of this application are to assess the usefulness of biomarkers, including p16 proteins, minichromosome maintenance (MCM) proteins, high-risk human papillomavirus (HPV) types, and E6 and E7 mRNA/oncoproteins, as adjunct tools to anal Pap smear in identifying HGAIN and to study the impact of HIV infection on the characteristics of anal cytology (by anal Pap smear) and biomarkers. To fulfill these goals, in addition to routine practice, it will be necessary to follow 450 MSM (315 HIV-positives and 135 HIV-negatives) over 60 months, and perform HRA and biomarkers on all clients at baseline and every 12 months. Information from this study would inform AIN screening and follow up approaches in HIV-positive and HIV-negative MSM in both resource-limited and resource-rich settings.

DETAILED DESCRIPTION:
The goals of this application are to assess the usefulness of biomarkers, including p16 proteins, MCM proteins, high-risk HPV types, and E6 and E7 mRNA/oncoproteins, as adjunct tools to anal Pap smear in identifying HGAIN and to study the impact of HIV infection on the characteristics of anal cytology (by anal Pap smear) and biomarkers. To fulfill these goals, in addition to routine practice, it will be necessary to follow 450 MSM (315 HIV-positives and 135 HIV-negatives) over 60 months, and perform HRA and biomarkers on all clients at baseline and every 12 months. Information from this study would inform AIN screening and follow up approaches in HIV-positive and HIV-negative MSM in both resource-limited and resource-rich settings.

ELIGIBILITY:
Inclusion Criteria:

* MSM with HIV negative
* MSM with HIV positive

Ages: 18 Years to 90 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: MSM with HIV negative and positive in Thailand
Sampling Method: Probability Sample
Enrollment: 450 (Actual)
Dates: Start 2009-12; Primary Completion 2015-08 (Actual); Study Completion 2017-05 (Actual)